CLINICAL TRIAL: NCT06210633
Title: XL STROKE: A Nationwide Prospective Registry of Endovascular Thrombectomy for Extra-large Ischemic Stroke With Large Vessel Occlusion
Brief Title: Prospective Registry of Endovascular Thrombectomy for eXtra-Large Ischemic Stroke
Acronym: XL-STROKE
Status: Recruiting | Type: Observational
Sponsor: Zhongming Qiu (Other)
Collaborators: Xiangtan Central Hospital (The Affiliated Hospital of Hunan University) (Unknown)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Other Study IDs: XL STROKE
Record Dates: First submitted 2024-01-05; First posted 2024-01-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke (AIS); Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: Acute ischemic stroke; large vessel occlusion; endovascular thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular thrombectomy: Patients in this group will be treated with medical management plus endovascular thrombectomy
  Interventions: Other: medical management; Other: endovascular thrombectomy
- Medical management: Patients in this group will be treated with guideline-based medical management alone
  Interventions: Other: medical management

INTERVENTIONS:
Other: medical management — Medical management will be based on the recommendations of the stroke management guidelines of the Chinese Stroke Association. Patients will receive intravenous thrombolysis according to the guidelines if they are eligible for thrombolysis. Patients who are not treated with intravenous thrombolysis will be treated with aspirin, unless an indication for early anticoagulation is present.
Other: endovascular thrombectomy — The use of devices (i.e. stent-retriever, aspiration catheter) is at the discretion of neurointerventionalist. Intra-arterial administration of alteplase, tenecteplase, tirofiban, angioplasty and stenting will also be permitted.
  Groups: Endovascular thrombectomy

SUMMARY:
Since 2015, many randomized trials have shown that endovascular thrombectomy improve functional outcomes in acute ischemic stroke patients with large vessel occlusion. Recently, five randomized controlled trials (ANGEL-ASPECT [Endovascular Therapy in Acute Anterior Circulation Large Vessel Occlusive Patients with a Large Infarct Core], LASTE [LArge Stroke Therapy Evaluation], RESCUE-Japan LIMIT [The Recovery by Endovascular Salvage for Cerebral Ultra-Acute Embolism-Japan Large Ischemic Core Trial], SELECT 2 [Randomized Controlled Trial to Optimize Patient's Selection for Endovascular Treatment in Acute Ischemic Stroke], and TENSION [The Efficacy and Safety of Thrombectomy in Stroke with extended lesion and extended time window]) demonstrated the efficacy and safety of thrombectomy for large infarct patients (defined as Alberta Stroke Program Early Computed Tomography Score [ASPECTS] ≥3 or infarct core <100ml). Patients with extra-large infarct core (ASPECTS score of 2 or less) were excluded from these trials. Therefore, the efficacy of endovascular thrombectomy in patients with extra-large ischemic burden has not been well studied. The XL STROKE registry is aiming to investigate the clinical outcomes and safety of mechanical thrombectomy in acute extra-large ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria

1. Age ≥18 years;
2. Presenting with acute ischemic stroke within 24 hours of time from last known well;
3. The patient or patient's representative signs a written informed consent form before enrollment.

Neuroimaging inclusion criteria

1. Occlusion of internal carotid artery, or the middle cerebral artery M1 or M2 segments confirmed by computed tomography angiography, magnetic resonance angiography, or digital subtraction angiography;
2. The baseline ASPECTS is 0 to 2 based on NCCT or diffusion weighted imaging, or cerebral extra-large ischemic core volume ≥85ml (defined as relative cerebral blood flow <30% on CT perfusion or an apparent diffusion coefficient <620×10^-6 mm2/s on MRI).

Exclusion criteria

1. CT or MRI evidence of acute intracranial hemorrhage;
2. Evidence of mass effect with ventricular effacement, midline shift or herniation on baseline imaging;
3. Females who are pregnant, or those of childbearing, potential with positive urine or serum beta Human Chorionic Gonadotropin test;
4. Previous bleeding disorders, severe heart, liver or kidney disease, or sepsis;
5. Any terminal illness with life expectancy less than 6 months;
6. Participation in other clinical treatment trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are presented with acute extra-large stroke and large vessel occlusion within 24 hours of time from last known well.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90±14 days after enrollment
  The primary outcome of this study is level of disability assessed by the score on the modified Rankin Scale at 90±14 days (scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death; mRS 6 and 5 will be merged as the worst outcome level to avoid a shift of 6 to 5 to be seen as better outcome).

SECONDARY OUTCOMES:
Independent ambulation | 90±14 days after enrollment
  Score of 0-3 on the modified Rankin scale
Not ambulatory nor capable of body self-care | 90±14 days after enrollment
  Score of 0-4 on the modified Rankin scale
Functional independence | 90±14 days after enrollment
  Score of 0-2 on the modified Rankin scale
Excellent outcome | 90±14 days after enrollment
  Score of 0-1 on the modified Rankin scale
National Institutes of Health Stroke Scale score | 5-7 days after enrollment or discharge (whichever occurred first)
  Scores on the National Institutes of Health Stroke Scale range from 0 to 42, with higher scores indicating worse neurologic deficits.
Health-related quality of life | 90±14 days after enrollment
  Health-related quality of life [European Quality Five-Dimension Five-Level (EQ-5D-5L) scale score]
Incidence of symptomatic intracranial hemorrhage | 48 hours after enrollment
  Use Heidelberg criteria to assess symptomatic intracranial hemorrhage.
Incidence of any intracranial hemorrhage | 48 hours after enrollment
  Any intracranial hemorrhage within 48 hours
Incidence of decompressive hemicraniectomy | 7 days after enrollment
  Decompressive hemicraniectomy during hospitalization
Mortality during hospitalization | 7 days after enrollment
  Death from any cause
Mortality | 90±14 days after enrollment
  Death from any cause
The occurrence of non-hemorrhagic serious adverse events | through study completion, an average of 90 days
  The occurrence of non-hemorrhagic serious adverse events, such as pneumonia, respiratory failure, circulatory failure, cerebral herniation, acute coronary syndrome, venous thrombosis.
Mortality within 1 year | One year after enrollment
  Death from any cause

OTHER OUTCOMES:
Modified Rankin Scale score at 1 year | One year after enrollment
  The score on the Modified Rankin Scale
Not ambulatory nor capable of body self-care | One year after enrollment
  Score of 0-4 on the modified Rankin scale
Independent ambulation | One year after enrollment
  Score of 0-3 on the modified Rankin scale
Functional independence | One year after enrollment
  Score of 0-2 on the modified Rankin scale
Excellent outcome | One year after enrollment
  Score of 0-1 on the modified Rankin scale
Health-related quality of life | One year after enrollment
  Health-related quality of life [European Quality Five-Dimension Five-Level (EQ-5D-5L) scale score]

CONTACTS AND LOCATIONS:
Overall Officials: Guangxiong Yuan, Principal Investigator — Xiangtan Central Hospital
Locations (1):
- Xiangtan Central Hospital, Xiangtan, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Clinical Study Report, and Analytic Code will be shared after approval of a proposal from principal investigator 3 years after the trial results are revealed.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 3 years after the trial results are revealed
Access Criteria: After approval of a proposal from principal investigator